CLINICAL TRIAL: NCT02732002
Title: Functional and Clinical Screening Assesment of the Shoulder Complex A New Methodological Model for Injury Management of Work Related Injuries
Brief Title: Functional and Clinical Screening Assesment of the Shoulder Complex A New Methodological Model for Injury Management
Acronym: FCSA
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Universidad Pública de Navarra (Other)
Collaborators: Mutua Navarra (Unknown)
Responsible Party: Principal Investigator, Dr Mikel Izquierdo, PhD, Universidad Pública de Navarra
Allocation: Not Applicable | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: MUT-001
Record Dates: First submitted 2016-04-02; First posted 2016-04-08 (Estimated); Last update posted 2016-04-08 (Estimated); Status verified 2016-04

CONDITIONS: Rotator Cuff Disease; Shoulder Impingement
Keywords: shoulder; rotator cuff- injury; management; rehabilitation model
MeSH Terms: conditions — Shoulder Impingement Syndrome; Rotator Cuff Injuries

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (1):
- OCBRA group. (Experimental): This group of patients will follow the proposed methodological approach for work related injuries rehabilitation.
  Interventions: Procedure: OCBRA ( Objective Criteria Based REhabilitation Algorithm

INTERVENTIONS:
Procedure: OCBRA ( Objective Criteria Based REhabilitation Algorithm — The patient will complete the initial functional and clinical evaluation in the medical room and laboratory. Afterwards, all the gathered information will be assembled to generate the patient-specific functional and clinical status-based rehabilitation program. This program will be generated in conjunction with the physical therapy staff. For each of the functional or clinical deficits observed during the examination, the physical therapist will identify the precise exercise and goal-based progression from a previously standardized goal-based rehabilitation algorithm adapted from previously published investigations targeting this issue

SUMMARY:
Work-related injuries of the shoulder complex represent a challenge for clinicians due to the large variety of clinical entities involved and the broad anatomic structures that are potentially affected. Furthermore, commonly performed orthopedic tests have demonstrated limited accuracy for the actual diagnosis of the injury. Although considerable research has been performed to standardize a model for shoulder injury management, a comprehensive approach integrating both a clinical and functional based status of the pathology and adapted rehabilitation prescription remains lacking.

The present study protocol aims to complement previously published shoulder injury management algorithms. Potentially, the multi-component, individualized and progressive multi-etiologic shoulder injury management model for rehabilitation could become a new effective strategy for reducing the time required to regain functional capacity and symptom recovery among patients with work-related shoulder injuries.

DETAILED DESCRIPTION:
The patient will be attended by an occupational physician who specializes in work-related injuries. Following medical diagnosis and supplementary evaluations where requested (i.e., radiological examination), the patient will be referred to the rehabilitation service. Before initiating the physiotherapeutic rehabilitation program, the patient will undergo a comprehensive functional screening at the biomechanics laboratory. Using a decision-making scheme, the identified functional deficits will be used to customize the individual rehabilitation plan.Registry procedures will be monitorized in a customized Microsoft excel spreadsheet which would record the code of patient episode (i.e. 20170001) as well as the number of the first medical and laboratory examination and the code of the therapist responsible of the rehabilitation. Twice a week an investigator (I.S) will check the report in order to assure proper patient rehabilitation course as well as claiming that pre and post laboratory and medical examinations are made. Completed episodes will be moved to another archive as "successfully completed" whereas in completed ones will be moved to another archive as "unsuccessfully completed". From that register efficacy data with regards to complete rehabilitation management model implementation rate will be calculated and reported apart from the outcome variables. The obtained results in terms of number of rehabilitation sessions performed and number of working day loss will be compared along with historical cohorts of the same medical institution

ELIGIBILITY:
Inclusion Criteria:

* Every Spanish speaking patient over 18 years of age and above the age of 64 seeking treatment by a physician at our institution due to work-related shoulder complaints from a mechanical origin (related to movement repetitions) lasting more than 4 weeks will be eligible to enter our rehabilitation model.

Exclusion Criteria:

* Shoulder pain episodes during less than 4 weeks. This preliminary time-based criterion for exclusion from the program is designed to prevent the inclusion of transient shoulder ailments that could adequately resolve with rest and AINES medication. This decision will prevent service saturation due to limited technical and human resources.
* Shoulder pain episodes corresponding to other shoulder pain sources other than work- related shoulder complaints from a mechanical origin

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 110 (Estimated)
Dates: Start 2016-09; Primary Completion 2017-09 (Estimated); Study Completion 2018-09 (Estimated)

PRIMARY OUTCOMES:
Pain | 1 year
  Pain levels during the complete clinical and functional examinations will be recorded using the previously validated Visual Analogue Score (VAS)
Active Range of Motion (AROM) | 1 year
  The shoulder range of motion (ROM) will be measured through the use of 3 iso-inertial unit STT-IBS (STT Systems, Spain) - based technology.
  The STT-IBS is a 9 degrees-of-freedom inertial measurement unit that integrates an accelerometer, a gyroscope and a magnetometer in each of its axes. The system measures the relative orientation, acceleration and position (in each of the X, Y, Z axes) of the STT-IBS sensors and sends this information to a computer with a Bluetooth-enabled host. The raw signals are processed online by iSens software (STT-Systems©, Spain), which provides the angular velocity, the acceleration and the angular position of each STT-IBS. Furthermore, after selecting the preferred model form the software (i.e., flexion/extension, FLX/EXT shoulder model) and placing the sensor units accordingly, the software provides the angular measurement of the selected movement in each plane.
Isometric Peak force evaluation | 1 year
  During the entire screening examination, each of the orthopedic tests performed will be performed with the implementation of a Hand-Held dynamometer (MicroFeet 1 Hoogan Industries, USA) to register the peak force (N) exerted during each task in addition to the standard clinical interpretation of the pain elicited during the maneuver. Routinely, 3 repetitions will be performed for each limb at each testing position. The first repetition will serve as familiarization, whereas the subsequent two repetitions will be registered for further analysis. The Orthopaedics test will include three different test for each of the examining clinical entity, such as shoulder impingement, instability, and weakness

SECONDARY OUTCOMES:
Measure of self reported shoulder function. Simple Shoulder Test Questionnaire (SST) | 1 year
  Self-reported shoulder function was registered by means of the utilization of the Simple Shoulder Test Questionnaire (SST). The questionnaire consists of 12 items, and dichotomous responses are registered (yes/no). Two questions are related to pain, 7 are related to function and strength and 3 are related to range of motion perceptions. The minimum clinically importance difference between pre- and post-rehabilitation evaluations was set between 2 to 2.33 points (Angst et al.2011)
Cost Effectiveness ratio | 1 year
  The economical burden of the rehabilitative process (by associating both medical and work missing economical costs) will be provided and compared to historical cohorts of the same medical institution (50 patients recruited the year before the OCBRA model is implemented) following the previously reported models (Goessens et al 2001J Clin Epidemiol)) . The number of overall rehabilitation and medical visitations made will by multiplied by its economical costs. The number of sessions administered as well as working day loss will be provided by hosting the Mutual Insurance society for work-related injury management. The economical burden of both medical and working day loss will be provided by the same institution following the recommendations of the National Social Health agency of the Spanish Heath Service Ministry. The cost effectiveness ratio will be calculated as the number of visitations made + working day loss divided by the sum of its economical burden

CONTACTS AND LOCATIONS:
Locations (1):
- Universidad Publica de Navarra, Tudela, Navarre, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] van der Heijden GJ. Shoulder disorders: a state-of-the-art review. Baillieres Best Pract Res Clin Rheumatol. 1999 Jun;13(2):287-309. doi: 10.1053/berh.1999.0021. PMID 10952865
- [Background] Larsson B, Sogaard K, Rosendal L. Work related neck-shoulder pain: a review on magnitude, risk factors, biochemical characteristics, clinical picture and preventive interventions. Best Pract Res Clin Rheumatol. 2007 Jun;21(3):447-63. doi: 10.1016/j.berh.2007.02.015. PMID 17602993
- [Background] van Rijn RM, Huisstede BM, Koes BW, Burdorf A. Associations between work-related factors and specific disorders of the shoulder--a systematic review of the literature. Scand J Work Environ Health. 2010 May;36(3):189-201. doi: 10.5271/sjweh.2895. Epub 2010 Jan 22. PMID 20094690
- [Background] Cools AM, Cambier D, Witvrouw EE. Screening the athlete's shoulder for impingement symptoms: a clinical reasoning algorithm for early detection of shoulder pathology. Br J Sports Med. 2008 Aug;42(8):628-35. doi: 10.1136/bjsm.2008.048074. Epub 2008 Jun 3. PMID 18523035
- [Result] Ginn KA, Cohen ML. Exercise therapy for shoulder pain aimed at restoring neuromuscular control: a randomized comparative clinical trial. J Rehabil Med. 2005 Mar;37(2):115-22. doi: 10.1080/16501970410023443. PMID 15788347
- [Result] Andersen LL, Fallentin N, Thorsen SV, Holtermann A. Physical workload and risk of long-term sickness absence in the general working population and among blue-collar workers: prospective cohort study with register follow-up. Occup Environ Med. 2016 Apr;73(4):246-53. doi: 10.1136/oemed-2015-103314. Epub 2016 Jan 6. PMID 26740688
- [Derived] Setuain I, Gonzalez-Izal M, Paularena A, Luque JL, Andersen LL, Izquierdo M. A protocol for a new methodological model for work-related shoulder complex injuries: From diagnosis to rehabilitation. BMC Musculoskelet Disord. 2017 Feb 7;18(1):70. doi: 10.1186/s12891-017-1435-2. PMID 28173784